CLINICAL TRIAL: NCT06029608
Title: Evaluation of the Efficacy and Safety of Magnetically-controlled Capsule Gastroscopy for Postoperative Assessment in Elderly Patients and Patients With Underlying Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaobo Li, Chief physician, Shanghai Jiao Tong University School of Medicine
Other Study IDs: Renji202302
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Evaluation,Efficacy,Safety
Keywords: Magnetically-controlled Capsule Endoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Magnetically-controlled Capsule endoscopy group: Using magnetic-controlled capsule gastroscopy for postoperative assessment in elderly patients and patients with underlying diseases
- Conventional endoscopy group: Using conventional endoscopy for postoperative assessment in elderly patients and patients with underlying diseases

SUMMARY:
The objective of this prospective, observational, controlled clinical study is to use magnetically-controlled capsule gastroscopy for postoperative assessment in elderly patients and patients with underlying diseases, to evaluate its clinical efficacy and safety.

DETAILED DESCRIPTION:
Gastric cancer is the most common digestive tract malignancy in China, which severely impacts human health and quality of life. Currently, surgery is the main treatment for gastric cancer. Since the surgery removes part or all of the stomach for malignant tumor, various postoperative complications inevitably occur. The occurrence of postoperative complications is detrimental to the prognosis of patients. Therefore, regular follow-up after surgery is necessary to closely monitor for upper gastrointestinal symptoms and periodically examine intragastric lesions in order to make timely diagnosis and treatment, and improve quality of life. Standard endoscopy procedures often cause discomfort and poor compliance in elderly patients. Also, for patients with severe respiratory diseases, severe cardiocerebral vascular diseases, the risks of anesthesia are extremely high. Magnetic-controlled capsule gastroscopy has the advantages of being completely painless, convenient, highly accurate in diagnosis, and well-accepted by patients. It is more suitable for postoperative assessment in elderly patients and patients with underlying diseases.

ELIGIBILITY:
Inclusion Criteria:

* Planned to undergo magnetic-controlled capsule gastroscopy or conventional endoscopy, and have undergone surgery for gastric malignant tumors (including surgical resection and ESD), elderly patients (older than 65 years) or patients with underlying diseases (cardiovascular, respiratory, hemorrhagic diseases, etc.);
* Agree to participate in this clinical trial and sign the informed consent form.

Exclusion Criteria:

* No surgical conditions or refuses abdominal surgery (Once the capsule is stuck it cannot be removed surgically);
* Cardiac pacemakers (except MRI-compatible ones);
* Electronic implants or metal foreign bodies;
* Pregnant women;
* Known or suspected GI obstruction, stenosis, fistula;
* Dysphagia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly patients (older than 65 years) and patients with underlying diseases (cardiovascular, respiratory, hemorrhagic diseases, etc.) who underwent surgery for gastric malignant tumors (including surgical resection and ESD).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-11-06 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Detection of gastric lesions (or postoperative complications) | 1 day
  Detection of gastric lesions (or postoperative complications)

SECONDARY OUTCOMES:
Upper gastrointestinal discomfort symptoms or not | 1 day
  Patients have or no upper gastrointestinal discomfort symptoms after surgery (such as nausea, vomiting, acid reflux, belching, bloating, postprandial fullness, and early satiety), judging by the patient's chief complaint.
Patients' comfort during the procedure | 1 day
  Use BCS to evaluate patients' comfort during the procedure (BCS is Bruggrmann comfort scale, a 5-point scale of 0 to 4, with a higher score indicating higher comfort.)
Gastric clarity and visibility | 1 day
  Assess the clarity and visibility of the stomach. The clarity and visibility of the field of vision is divided into three categories, that is, class I: the field of vision is clear, and the part and mucosa can be accurately observed; Class II: Vision is not clear, but can still distinguish the part; Class III: Cloudy vision, unable to distinguish the area.
Detection of small intestinal and colonic lesions in the magnetic-controlled capsule endoscopy group | 1 day
  Detection of small intestinal and colonic lesions in the magnetic-controlled capsule endoscopy group

CONTACTS AND LOCATIONS:
Locations (1):
- Departments of Gastroenterology and Clinical Laboratory, Shanghai Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No